CLINICAL TRIAL: NCT05416203
Title: Brief Enhanced Anxiety Sensitivity Treatment: A Pilot Study
Brief Title: BEAST: A Pilot Trial
Acronym: BEAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3880-P; I02RX003880 (Other Grant/Funding Number: VA RR&D); NCT05490199 (obsolete NCT alias)
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Anxiety Sensitivity; Functional Impairment
Keywords: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants will all be enrolled to receive the active intervention, Brief Enhanced Anxiety Sensitivity Treatment.
Masking Description: No masking will occur as this is a one-arm trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BEAST Condition (Experimental): A one-session intervention that can be delivered effectively by a clinician via telehealth and supplemented with a mobile app to provide opportunities to practice the skills learned in the face-to-face session.
  Interventions: Behavioral: Brief Enhanced Anxiety Sensitivity Treatment

INTERVENTIONS:
Behavioral: Brief Enhanced Anxiety Sensitivity Treatment — BEAST is a CBT-based intervention that includes psychoeducation, identifying and challenging maladaptive thoughts, and interoceptive exposure. The intervention is delivered through a single virtual face-to-face session supplemented with a mobile app for two weeks after the face to face session.
  Other Names: BEAST

SUMMARY:
This pilot study trial will test the acceptability, feasibility, and usability of a brief enhanced anxiety sensitivity treatment to reduce anxiety sensitivity and functional impairment in Veterans.

DETAILED DESCRIPTION:
This study tests a treatment with two components: first, there is a single session face-to-face virtual intervention delivered by the counselor or therapist via VA Video Connect software. Second, a mobile app (mPRO) is used for EMA and to deliver EMI components.

Veterans will be enrolled following informed consent. The research staff will read the measures to the Veteran who will verbally provide their answers.

Veterans will next complete the baseline assessment. At the baseline assessment, Veterans meet with the Project Coordinator by phone or virtually to complete a consenting process, guidance on the video software being used, and set-up and guidance on use of the mobile app.

Following the baseline assessment, participants will be scheduled to receive the face-to-face virtual intervention followed by two weeks of EMA/EMI via mPRO.

At the end of the two weeks, Veterans will complete a post-intervention assessment appointment. The post-intervention assessment includes an exit interview for participants to provide additional feedback regarding acceptability of the intervention.

Follow-up assessment appointments will be completed at the 1-month and 3-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Are English-speaking
* Score equal to or greater than 9 on the SSASI indicating elevated anxiety sensitivity
* Score equal to or greater than 5 on the WHODAS 2.0

Exclusion Criteria:

* Veterans with cognitive impairment as measured scoring equal to or greater than 11 on the Blessed
* Orientation-Memory-Concentration Test
* Veterans without access to a smartphone
* Veterans with significant medical or psychiatric conditions that may limit participation, including:

  * severe documented schizophrenia
  * an ongoing active psychotic or manic state
  * an imminent suicide crisis will be excluded from our study and provided the appropriate referral

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas P Allan, PhD, Principal Investigator — VA Finger Lakes Healthcare System, Canandaigua, NY
Locations (1):
- VA Finger Lakes Healthcare System, Canandaigua, NY, Canandaigua, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BEAST Condition
Started | 15
Completed Intervention | 14
Completed | 13
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | BEAST Condition
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.87 (5.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
Marital Status [Count of Participants; unit: Participants]
  Single/Never Married | 4
  Divorced/Separated | 4
  Married or Living with Partner | 7
Education [Count of Participants; unit: Participants]
  High School Diploma | 3
  Associates/Technical | 3
  Four-Year College | 3
  Master's Degree | 5
  Professional Degree | 1
Served During Gulf War [Count of Participants; unit: Participants]
  Served during Gulf War | 6
  Did not Serve during Gulf War | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Anxiety Sensitivity
Description: Anxiety sensitivity will be measured via the Anxiety Sensitivity Index-3, an 18-item self-report measure assessing fear of negative consequences of anxiety-related symptoms. Scores range from 0 to 72 with higher scores indicating worse anxiety sensitivity.
Time Frame: From baseline to post-intervention (two-weeks after virtual treatment session)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BEAST Condition
Number analyzed (Participants) | 13
score on a scale | -11.15 (13.89)

2. Primary Outcome: Program Satisfaction
Description: Program satisfaction will be measured using an adapted 11-item version of the Program Satisfaction Questionnaire that assesses both general program satisfaction (usefulness, acceptability) and perceived utility of program components (psychoeducation, EMA/EMI schedule). Average scores range from 1 to 5 with higher scores indicating greater satisfaction.
Time Frame: Post-intervention (two weeks after virtual treatment session)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- BEAST Condition: A one-session intervention that can be delivered effectively by a clinician via telehealth and supplemented with a mobile app to provide opportunities to practice the skills learned in the face-to-face session.
  Brief Enhanced Anxiety Sensitivity Treatment: BEAST is a CBT-based intervention that includes psychoeducation, identifying and challenging maladaptive thoughts, and interoceptive exposure. The intervention is delivered through a single virtual face-to-face session supplemented with a mobile app for two weeks after the face to face session. The average score ranges from 1 to 5 with higher scores indicating greater satisfaction.
Arm/Group | BEAST Condition
Number analyzed (Participants) | 13
score on a scale | 3.95 (.77)

3. Primary Outcome: Mean Change in Functional Impairment
Description: Functional impairment will be measured using the 12-item version of the World Health Organization Disability Assessment 2.0. This scale assesses functional impairment across six domains: 1) understanding and communication, 2) self-care, 3) mobility, 4) interpersonal relationships, 5) work and household roles, and 6) community and civic roles. Scores range from 0 to 48 with higher scores indicating worse functional impairment.
Time Frame: From baseline to post-intervention (two-weeks after virtual treatment session)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BEAST Condition
Number analyzed (Participants) | 13
score on a scale | -7.38 (10.94)

4. Secondary Outcome: Mean Changes in Anxiety
Description: Changes in anxiety will be measured using the 8-item PROMIS anxiety short form. Scores range from 8 to 40 with higher scores indicating worse outcome.
Time Frame: From baseline to follow-up (measured six weeks after intervention session)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BEAST Condition
Number analyzed (Participants) | 13
score on a scale | -6.62 (8.42)

5. Secondary Outcome: Mean Changes in Worry Related to the COVID-19 Pandemic
Description: Worry related to the pandemic will be measured using the Coronavirus Impact Battery - Worry Scale. This scale is an 11-item scale measuring distress and worry due to the COVID-19 pandemic. Scores range from 0 to 44 with higher scores indicating worse outcome.
Time Frame: From baseline to follow-up (measured six weeks after intervention session)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BEAST Condition
Number analyzed (Participants) | 13
score on a scale | -9.67 (13.34)

6. Secondary Outcome: Mean Changes in Avoidance Due to the COVID-19 Pandemic
Description: Avoidance due to the pandemic will be measured using the Coronavirus Impact Battery - Behavior Scales, a 12-item scale assessing avoidance behaviors in relation to the COVID-19 pandemic. Scores range from 0 to 48 with higher scores indicating worse outcome.
Time Frame: From baseline to follow-up (measured six weeks after intervention session)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BEAST Condition
Number analyzed (Participants) | 13
score on a scale | -.15 (8.51)

7. Secondary Outcome: Mean Changes in Functional Impairment Due to the COVID-19 Pandemic
Description: Functional Impairment Due to COVID ScaleA 7-item measure adapted from the WHODAS 2.0 to capture difficulties in functioning due to the COVID-19 pandemic. Scores range from 0 to 28 with higher scores indicating worse outcomes.
Time Frame: From baseline to follow-up (measured six weeks after intervention session)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BEAST Condition
Number analyzed (Participants) | 13
score on a scale | -1.58 (4.50)

8. Secondary Outcome: Mean Change in Depression
Description: Changes in depression will be measured using the 4-item depression scale from the PROMIS Profile-29. The scores range from 4-20 with higher scores indicating worse outcomes.
Time Frame: From baseline to follow-up (measured six weeks after intervention session)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BEAST Condition
Number analyzed (Participants) | 13
score on a scale | -2.92 (2.72)

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Arm/Group | BEAST Condition
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT05416203/Prot_SAP_001.pdf
  • Informed Consent Form (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/03/NCT05416203/ICF_000.pdf